CLINICAL TRIAL: NCT07355829
Title: DemTool - Supporting Life With Dementia
Acronym: DemTool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Dementia Research Centre (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DemTool
Record Dates: First submitted 2025-12-10; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dementia (Diagnosis)
Keywords: Family caregivers; dementia; Psychosocial intervention
MeSH Terms: conditions — Dementia; Disease | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The trial included 15 municipalities in the intervention group. Family caregivers in the intervention group received one or two of the tailored interventions based on their level of burden and specific needs, as assessed by the local primary care dementia coordinator in the municipality. The interventions included: 1) a support group focused on addressing caregiver burden, providing both professional and peer support; 2) a group course consisting of six sessions aimed at helping caregivers cope with everyday challenges; and 3) a group course over five sessions that offered information on dementia, transitioning to a nursing home, person-centered care, and effective communication strategies.
  Interventions: Behavioral: Life with dementia in the community - Support group for family caregivers; Behavioral: Life with dementia in the community - Group course; Behavioral: Life with dementia in a care home- Group course
- Treatment-as-usual (No Intervention): The trial included 15 municipalities in the treatment-as-usual group. Family caregivers in the treatment-as-usual group had access to local health and social services in their municipality, including support and information from primary care dementia coordinators, support groups, hotlines provided by patient associations, and respite care for the person with dementia in a home or daycare setting.

INTERVENTIONS:
Behavioral: Life with dementia in the community - Support group for family caregivers — This intervention aimed to promote coping and reduce caregiver burden through professional and peer support. It was delivered over a varied number of sessions, as this depended on the number of recruited participants in the municipalities. To support these sessions, booklets and fact sheets for family caregivers could be incorporated. These materials would cover various topics, including the psychological challenges and reactions faced by family caregivers, guidance on effective communication with people with dementia, and a guide to practical and legal issues. Further, there would be fact sheets addressing specific symptoms, such as memory loss, communication difficulties, depression, apathy, behavioral changes, and reduced awareness of symptoms. The use of these booklets and fact sheets in the intervention would be determined by the municipalities, allowing for adaptation to fit local contexts. Dementia coordinators within the community setting would implement this intervention.
  Arms: Intervention
Behavioral: Life with dementia in the community - Group course — This intervention aimed to provide information on, e.g., dementia diseases, everyday life with dementia, being a family caregiver, and planning the future. It was delivered over six sessions. To support the sessions, booklets and fact sheets for family caregivers were incorporated. Materials covered various topics, including, e.g., the psychological challenges and reactions faced by family caregivers, and information on accessing support and services. Additionally, fact sheets addressed specific symptoms, such as memory loss, communication difficulties, apathy, and behavioral changes. To support municipalities in implementing this intervention, the Danish Dementia Research Centre provided PowerPoint presentations and a suggested order for the topics covered in each session. However, municipalities have the flexibility to adapt the use of the PowerPoints and the sequence of the sessions to suit their local contexts. This was done by dementia coordinators within the community setting.
  Arms: Intervention
Behavioral: Life with dementia in a care home- Group course — This intervention aimed to provide information on dementia diseases, moving into a care home, person centered care, and communication. It was delivered over five sessions. To support the sessions, booklets and fact sheets for family caregivers were incorporated. Materials covered various topics, including, e.g., psychological challenges and reactions faced by family caregivers, and guidance on effective communication with people with dementia. Additionally, fact sheets addressed specific symptoms, such as memory loss, communication difficulties, behavioral changes, and reduced awareness of symptoms. To support municipalities in implementing this, the Danish Dementia Research Centre provided PowerPoint presentations and a suggested order for the topics covered in each session. However, municipalities have the flexibility to adapt the use of PowerPoints and the sequence of sessions to suit their local contexts. This was carried out by dementia coordinators within the community setting.
  Arms: Intervention

SUMMARY:
This study will investigate the effects of a Danish psychosocial intervention, specifically the DemTool - supporting life with dementia, on quality of life and caregiver strain in family caregivers of people with dementia.

DETAILED DESCRIPTION:
'DemTool - supporting life with dementia' was developed in Denmark by the Danish Dementia Research Centre with a focus on improving the quality of life of people with dementia and their family caregivers. DemTool was developed to assist professional caregivers in Danish municipalities. It is intended for use by professionals responsible for counseling and educating patients and their family caregivers in primary care settings. This study will examine the impact of DemTool on the quality of life and caregiver strain among family caregivers of individuals with dementia using self-reported data from questionnaires. Family caregivers who participated in the intervention were invited to complete a questionnaire before their inclusion in the study, which served as a baseline measure. They then filled out a follow-up questionnaire approximately one month after receiving their last intervention. Meanwhile, the treatment-as-usual group also completed a questionnaire before study inclusion and received a follow-up questionnaire two months after the baseline measure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at enrollment.
* Providing care for a family member with dementia.
* Speaking and understanding Danish.

Exclusion Criteria:

* Unable to give informed consent for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Neuropsychiatric Inventory - Distress (NPI-D) | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  Used to measure the emotional and psychological burden experienced by caregivers of patients with dementia.
Change from baseline in European Quality of Life-Visual Analogue Scale (EQ VAS). | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  Used to measure a person's self-assessed general health on a given day. It's a vertical line scale from 0 (worst imaginable health) to 100 (best imaginable health), where respondents mark their current health state.

SECONDARY OUTCOMES:
Change from baseline in the 5-level EQ-5D version (EQ-5D-5L). | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  Used to measure quality of life in five dimensions, on a 5-point likert scale. Completing it generates a one-digit number for each dimension, which can be converted into a utility score. The closer the utility value is to 1, the better the health state. The EQ-5D-5L utility ranges from -0.757 to 1.
Change from baseline in World Health Organization Wellbeing Index (WHO-5). | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  Assesses subjective psychological well-being over the past two weeks. Five questions are rated on a 6-point Likert scale. A higher score indicates better wellbeing.
Change from baseline in University of California, Los Angeles Three-Item Loneliness Scale (UCLA 3-item). | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  Used to assess feelings of loneliness or social isolation via three questions on relational and social connectedness, and self-perceived isolation, rated on a 3-point Likert scale. Higher scores reflect greater loneliness.
Change from baseline in Carer Experience Scale (CES). | Outcome were measured at baseline (study inclusion) and follow-up (1 month after the last received intervention and 2 months from baseline in the treatment-as-usual group).
  A measure of caregiving experience in everyday life operationalized in six questions on a 3-point Likert scale. A total index score, calculated by adding preference weights, ranges from 0 to 100, where 0 indicates the poorest and 100 the best caregiving experience.

CONTACTS AND LOCATIONS:
Overall Officials: Gunhild Waldemar, MD, D.M.Sc, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark.; T. Rune Nielsen, PhD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark.; Ann Nielsen, MSPH, PhD, Principal Investigator — Danish Dementia Research Centre, Rigshospitalet, Copenhagen, Denmark.
Locations (1):
- Danish Dementia Research Centre, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
While the study data are pseudonymized, participants did not consent to have their data shared with third parties beyond the study team. The informed consent form clearly restricted data usage to analyses conducted within the project and the publication of aggregated results in scientific articles. Sharing individual-level data would go beyond the original consent. Therefore, the dataset cannot be made publicly available.